CLINICAL TRIAL: NCT05743452
Title: Clinical Trial on the Safety and Efficacy of Magnesium Doped Calcium Silicate 3d Alveolar Bone Repair Unit for Periodontal Bone Defects
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0535
Record Dates: First submitted 2023-02-05; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Device: GBR with CS@Mg The patient was treated by GBR with magnesium calcium silicate scaffold for alveolar bone defect.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS@Mg (Experimental): The patient was treated by GBR with magnesium calcium silicate scaffold for alveolar bone defect.
  Interventions: Device: GBR with CS@Mg

INTERVENTIONS:
Device: GBR with CS@Mg — The patient was treated by GBR with magnesium calcium silicate scaffold for alveolar bone defect.

SUMMARY:
The goal of this clinical trial is to test in height increment of alveolar bone and safety evaluation index.

The main question it aims to answer are:

• The safety and effectiveness of magnesium calcium silicate three-dimensional alveolar bone repair unit in the repair of periodontal bone defects Participants will be treated through Guided Bone Regeneration operation with calcium magnesium silicate three-dimensional alveolar bone repair unit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old, healthy;
* Good oral hygiene, do not smoke;
* There is bone defect at the tooth extraction site, and it is planned to carry out implant repair after tooth extraction;
* There is at least one healthy adjacent tooth in the mesial and distal surface of the tooth extraction site;
* The residual height from the bottom of the extraction socket to the crest of the alveolar ridge is ≥ 3 mm, with at least one bone wall;
* Can understand the purpose of the trial
* Be willing to cooperate with surgical treatment and follow-up, voluntarily participate in the trial
* Sign the informed consent form.

Exclusion Criteria:

* The affected tooth is in the acute inflammatory stage;
* Those who have bad habits such as smoking and drinking；
* Subjects who cause artifacts in oral imaging examination, such as the extraction site and its adjacent teeth are metal Dentures, porcelain teeth;
* Patients are allergic to ceramic implants;
* Those who have participated in other clinical trials in the past 3 months;
* The investigator estimated that the compliance was poor, or there were other factors that were not suitable for the test;
* Patients with a history of diabetes or abnormal blood glucose detection (fasting blood glucose ≥ 7mmol/L);
* Abnormal liver and kidney function (AST, ALT, creatinine ≥ 1.5 times ULN);
* Patients with serious endocrine and metabolic diseases;
* Have a history of tertiary hypertension;
* Have a history of osteoporosis;
* Those who are not suitable for surgery due to the history of malignant tumor or other serious diseases;
* People with a history of autoimmune diseases;
* Pregnant or lactating women;
* Mental disorders without autonomous behavior ability;
* Patients who are using steroids that interfere with calcium metabolism within 3 months before the signing of informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Horizontal bone width | 24 weeks after operation
  The width of buccal lingual alveolar ridge was measured 1 mm below the crest of alveolar ridge.
Evaluation of wound healing | 2 weeks after operation
  The wound healing evaluation scale was modified according to the indicators described by Lobene et al (1986) and will be used to evaluate the wound healing after surgery. The gingival tissue in the material implantation area was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral Medicine, the Second Affiliated Hospital School of Medicine of Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No